CLINICAL TRIAL: NCT05185466
Title: The Effect of Nurse-Supported Self Management Programme on the Sustained Attention and Sleep Quality of the Nurses Working at Night Shift
Brief Title: Self Management Programme on the Sustained Attention and Sleep Quality of the Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Merve Çolak, Teaching Assistant, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 61351342/Ocak 2021-88
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Sleep Quality; Attention; Nurses
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group
  Interventions: Behavioral: Nurse-Supported Self Management Programme
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Behavioral: Nurse-Supported Self Management Programme — Training and incentives to improve nutrition habits and sleep health.
  Arms: Experimental Group

SUMMARY:
The aim of this study is to examine the effect of the nurse-supported self-management program on the sustained attention and sleep quality of night shift nurses. The self-management program consists of training and incentives for night shift nurses to gain healthy eating habits and improve their sleep health.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in shifts
* Those between the ages of 18-65
* Those who agree to participate in the study.

Exclusion Criteria:

* Pregnant and having suspicion of pregnancy
* Having vision and hearing problems
* Having diagnosed sleep disorder
* Having a chronic disease that will prevent participation in the study
* Having a diagnosed mental health problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-01-07 (Estimated); Study Completion 2022-03-07 (Estimated)

PRIMARY OUTCOMES:
Sustained Attention | First Month
  Psychomotor Vigilance Test
Sleep Quality | First Month
  Pittsburgh Sleep Quality Index (PSQI)
Sleepiness | First Month
  Epworth Sleepiness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Merve Çolak, MSc, Principal Investigator — T.C. Üsküdar Üniversitesi
Locations (1):
- Istanbul / Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colak M, Esin MN. The Effect of Nurse-Led Self-Management Program on Psychomotor Vigilance and Sleep of Nurses Working Night Shifts: A Randomised Controlled Trial. Int J Nurs Pract. 2025 Dec;31(6):e70076. doi: 10.1111/ijn.70076. PMID 41188198